CLINICAL TRIAL: NCT05038085
Title: The Effect of Health Education and Progressive Muscle Relaxation Exercise Program Applied Online on Postpartum Depression and Maternal Attachment: a Randomized Controlled Study
Brief Title: Postpartum Depression and Maternal Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Canan Uçakçı Asalıoğlu, research asistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021 - 175
Record Dates: First submitted 2021-07-16; First posted 2021-09-08 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Depression; Progressive Muscle Relaxation
Keywords: postpartum depression; maternal attachment; progressive muscle relaxation exercise; online health education
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: parallel randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group application (Experimental): progressive muscle relaxation exercise health education
  Interventions: Behavioral: progressive muscle relaxation exercise
- control group application (No Intervention): No intervention will be made in the control group.

INTERVENTIONS:
Behavioral: progressive muscle relaxation exercise — 36-37 with pregnant women in the experimental group. There will be two online interviews starting from week one. Before the first interview, the PMRE video will be sent to the women, explained by the researcher. In the first meeting, basic information about postpartum depression and what to do to prevent postpartum depression and its treatment will be explained. The women will then be asked to describe the PKGE. "Relaxation Exercises CD Audio Recordings" belonging to the Turkish Psychological Association will be sent to women, and they will be asked to perform PMRE at least 3 days a week until delivery, accompanied by the instructions on the CD. In the second meeting; maternal attachment will be explained. In this interview, women will be asked to continue to do PMRE at least 3 days a week from the day they feel ready, starting at the latest 1 week after delivery.
  Other Names: health education
  Arms: experimental group application

SUMMARY:
In terms of postpartum care and depression, follow-up and controls should be continued online in order not to interrupt the follow-up and treatment of women. In this context, in order to prevent the development of postpartum depression and to increase maternal attachment, it is planned to deliver the progressive muscle relaxation exercise and individual health education program that we planned in our study through online applications. This study will be conducted to evaluate the effect of online health education and progressive muscle relaxation exercise program on postpartum depression and maternal attachment.The study was planned as a parallel randomized controlled experimental study conducted in a Family Health Center in Ankara, with a single-center, stratified block randomization (parity: primiparous, multiparous; EPDS score: 0-9, 10-30).The number of pregnant women to be included in the study was calculated as 56.Personal Information Form, Prenatal Attachment Scale, Edinburgh Postpartum Depression Scale and Postpartum Attachment Scale will be used to collect data.

DETAILED DESCRIPTION:
Sample Power analysis was performed to determine the number of samples. For this, the information in a similar study (Aydın Özkan et al., 2020) was used as a reference. The minimum number of participants required to be included in each group was determined as 24, with a total of 48 (α=0.01, 1-β=0.95). However, considering the loss rate (18.75%) in Aydın Özkan's study, which was taken as a reference, the total number of participants was determined as 56 (experimental: 28, control: 28).

Randomization In order to prevent imbalance between the groups, pregnant women will be assigned to the experimental and control groups by the tanned block randomization method. Pregnant women will be stratified according to parity (primiparous-multiparous) and Edinburgh Postpartum Depression Scale score (0-9 points, 10-30 points). In this context, 8 groups will be formed as shown below.

Set 1: Primiparous and pregnant women with EPDS scores between 0 and 9 Set 2: Primiparous and pregnant women with a EPDS score of 10-30 Set 3: Multiparous and pregnant women with EPDS score between 0 and 9 Set 4: Multiparous and pregnant women with a EPDS score of 10-30 Data Collection Personal Information Form, Prenatal Attachment Scale, Edinburgh Postpartum Depression Scale and Postpartum Attachment Scale will be used to collect data.

The purpose and content of the study will be explained by interviewing 35-week-old pregnant women who applied to FHCs for pregnancy follow-up. Their compliance with the sampling inclusion criteria will be evaluated. Then, an informed consent form will be signed by the pregnant women who agree to take part in the study. Personal information form, Prenatal Attachment Scale and Edinburgh Postpartum Depression Scale will be administered to pregnant women participating in the research. Then, the pregnant women will be randomized by stratified blocking according to their parity and EPDS score averages, and the assignment of the experimental and control groups will be made. Contact information (Phone numbers and e-mail addresses) will be taken at the first encounter.Experimental Group Application 36-37 with pregnant women in the experimental group. There will be a total of two online interviews, once a week, starting from the first week. Before the first interview, women will be sent a PKGE video explained by the researcher via e-mail or Whatsapp application, and they will be asked to watch it before the interview. In the first meeting, basic information about postpartum depression and what to do to prevent postpartum depression will be explained. The women will then be asked to describe the PKGE. The interview will be terminated when it is confirmed that the women have understood correctly and fully. Afterwards, "Relaxation Exercises CD Audio Recordings" belonging to the Turkish Psychological Association will be sent to the women, and they will be asked to do PCGE at least 3 days a week until delivery, accompanied by the instructions on the CD. In the second meeting; If postpartum depression develops, what should be done and maternal attachment will be explained, and women's opinions and questions about PCGE will be taken. In this interview, women will be asked to continue PCGE at least 3 days a week from the day they feel ready, starting at the latest 1 week after delivery.

During the application process to women, "Don't forget to do your relaxation exercise" every other day, "Weekdays to talk to your nurse about the training issues you have received. Weekend …. You can call or send a message about the issues you want to consult between the hours of the day. message will be sent. If the woman wants to have an interview, she will be called at the specified times and interviewed and the participant's questions will be answered. If it is noticed that an issue that needs help from different disciplines or that a postpartum complication develops, he will be referred to the hospital.

The Edinburgh Postpartum Depression Scale and the Postpartum Attachment Scale will be administered at the sixth week postpartum. The scales will be converted into an online questionnaire and mothers will be asked to fill in by sending their contact address.

Control group application Prenatal Attachment Scale and Edinburgh Postpartum Depression Scale will be administered to women at 35 weeks of pregnancy, Postpartum Attachment Scale and Edinburgh Postpartum Depression Scale will be administered to women at 6 weeks postpartum. The scales will be converted into an online questionnaire and women will be asked to fill in by sending their transportation address. No intervention will be applied to the women in the control group during the study.

ELIGIBILITY:
Inclusion Criteria:

* Being at least literate
* Being at least 18-35 years old
* Being between 35-36 weeks of pregnancy
* Not having any psychiatric diagnosis
* Not being pregnant at risk
* Being pregnant naturally
* Having the technical means to use Whatsapp® application
* Volunteering to participate in the research
* Not having a communication barrier

Exclusion Criteria:

* Having a stillbirth
* Hospitalization of the newborn
* Hospitalization of the mother
* The woman's desire to leave the research
* Not filling out data collection tools
* Unable to reach for training/consulting
* The woman's progressive relaxation exercise less than three days a week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The Edinburgh Postpartum Depression Scale (EPDS), Prenatal Attachment Scale (PAS) | prenatal 35. week
  PAS and EPDS will be administered to women at 35 weeks of pregnancy.The scales will be converted into an online questionnaire and mothers will be asked to fill in by sending their contact address.
  The lowest score that can be obtained from EPDS is 0 and the highest score is 30.Women with a total scale score higher than the cut-off point are considered to be a risk group in terms of postpartum depression.A minimum of 21 points and a maximum of 84 points can be obtained from the PBE. The increase in the score obtained by the pregnant indicates that the level of attachment also increases.

SECONDARY OUTCOMES:
The EPDS, The Postpartum Attachment Scale (PPAS) | postpartum 6. week
  The EPDS and the PPAS will be administered at the sixth week postpartum. The scales will be converted into an online questionnaire and mothers will be asked to fill in by sending their contact address.The lowest score that can be obtained from EPDS is 0 and the highest score is 30.Women with a total scale score higher than the cut-off point are considered to be a risk group in terms of postpartum depression.The cut-off point for PPAS is 26 points. A score of 27 or more from the overall scale is defined as having a postpartum attachment problem.

CONTACTS AND LOCATIONS:
Overall Officials: Şengül Yaman Sözbir, Assoc., Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No